CLINICAL TRIAL: NCT03123367
Title: An Evaluation of the Safety and TechnIcal Feasibility Of the NelLa Women's Care Line for Female Gynecological ExaminaTions and Procedures (VIOLET)
Brief Title: Evaluation of the Nella Women's Care Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceek Enterprises (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLP-0001
Record Dates: First submitted 2017-03-05; First posted 2017-04-21 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Group 1: Nella VuSleeve (Active Comparator): Sleeve
  Interventions: Device: Group 1: Nella VuSleeve
- Group 2: Nella NuSpec (Active Comparator): Speculum
  Interventions: Device: Group 2: Nella NuSpec
- Group 3: NellaSpec (Active Comparator): Speculum
  Interventions: Device: Group 3: NellaSpec
- Group 4: Nella Insert (Active Comparator): Sleeve
  Interventions: Device: Group 4: Nella Insert

INTERVENTIONS:
Device: Group 1: Nella VuSleeve — Sleeve
  Arms: Group 1: Nella VuSleeve
Device: Group 2: Nella NuSpec — Speculum
  Arms: Group 2: Nella NuSpec
Device: Group 3: NellaSpec — Speculum
  Arms: Group 3: NellaSpec
Device: Group 4: Nella Insert — Sleeve
  Arms: Group 4: Nella Insert

SUMMARY:
Evaluation of the Nella Women's Care Line

DETAILED DESCRIPTION:
The Nella Women's Care Line is being studied in women undergoing a gynecological exam and other gynecological procedures that require visibility and access to the cervix.

ELIGIBILITY:
General inclusion criteria (applies to all study groups):

* Subject is female
* Subject is 18 - 65 years of age, inclusive, at the time of consent
* Subject is undergoing a gynecological examination (as defined above) as part of their regular clinical care
* Subject has undergone one or more prior gynecological exams
* Subject is willing and able to provide written informed consent
* Subject is able and willing to perform the functions required by the study protocol

General exclusion criteria (applies to all study groups):

* Subject has undergone hysterectomy
* Subject has a known history of allergies to latex or plastics
* Subject is pregnant
* Subject is post-partum (≤ 12 weeks)
* Subject has had an induced or spontaneous abortion in the prior 12 weeks
* Subject has an active gynecologic complaint that, in the opinion of the clinician, would confound study results
* Subject has dyspareunia
* Subject has a known history of vulvodynia such as vulvular vestibular syndrome
* Subject has a known history of vaginismus
* Subject has a planned surgical procedure along with the gynecological exam
* Subject is under incarceration
* Subject is unable to provide written informed consent

Device specific inclusion criteria:

In addition to the general inclusion, the subject must meet all device specific criteria associated with their assignment group. Below are device-specific criteria. There is no device-specific exclusion criterion.

Nella VuSleeve (Group 1) inclusion:

• Subject has a BMI ≥ 30 and/or 3 or more vaginal births

NellaSpec (Group 2), Nella NuSpec (Group 3), and Nella Insert (Group 4) inclusion:

• Subject has a BMI < 35

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 154 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Technical Feasibility | Day of Exam or Procedure
  Cervical visualization and access

SECONDARY OUTCOMES:
Safety | Day of Exam or Procedure
  Number of Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Ceek Clinical Research, Study Director — Ceek Enterprises
Locations (1):
- Research Site, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided